CLINICAL TRIAL: NCT07086703
Title: Targeted Temperature Management at 33°C Versus Controlled Normothermia for In-hospital Cardiac Arrest
Acronym: IH-TTM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC23_0488
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induced hypothermia at 33°C: (Experimental)
  Interventions: Other: Induced hypothermia at 33°C
- Control normothermia (Active Comparator)
  Interventions: Other: Control normothermia

INTERVENTIONS:
Other: Induced hypothermia at 33°C — Cooling and maintenance phase :
  The aim is to achieve the target temperature of 33±0.5°C within 60 minutes after randomization. The target temperature of 33±0.5°C and device setting of 33°C will be maintained until 28 hours after randomization.
  - Rewarming: Normothermia will be restored by gradual rewarming at a rate of 0.2°C/h.
  - After rewarming: After 40 hours, in those participants who are still comatose or sedated, normothermia (36.5-37.7°C) will be maintained until 72 hours after randomization, and active warming will be avoided.
  Arms: Induced hypothermia at 33°C:
Other: Control normothermia — Participants whose initial temperature is below 33°C may be actively rewarmed to 36.5°-37.7°C, at which point active rewarming will be stopped and passive rewarming performed according to the latest guidelines. Participants whose initial temperature is above 33°C will not be actively rewarmed to normothermia. The goal will be to maintain temperature no higher than 37.8°C.
  After 40 hours, in those participants who are still comatose or sedated, normothermia (36.5-37.7°C) will be maintained until 72 hours after randomization, and active warming will be avoided.
  Arms: Control normothermia

SUMMARY:
The IH-TTM trial is designed to determine whether survival with a favorable neurological outcome is improved by induced hypothermia at 33°C in comatose critically ill patients admitted after resuscitated in-hospital cardiac arrest (IHCA). Recent evidence suggests that targeted temperature management (TTM) at 33°C may provide no survival benefits compared to controlled normothermia in unselected patients with out-of-hospital cardiac arrest (OHCA). However, this evidence is relevant only to OHCA of presumed cardiac origin, chiefly witnessed and immediately followed by resuscitation efforts. Only scant data are available for cardiac arrest (CA) of other origins and for IHCA.

In a randomized clinical trial of patients with CA in an initial non-shockable rhythm, the subgroup with IHCA had significantly better outcomes when treated with TTM at 33°C versus controlled normothermia; nevertheless, the sample size was limited. Another randomized controlled trial done specifically in patients with IHCA failed to show benefits of TTM at 33°C compared to controlled normothermia but was underpowered. Thus, whether therapeutic hypothermia is indicated after IHCA remains unclear. IH-TTM will be the largest trial assessing TTM after IHCA.

ELIGIBILITY:
Inclusion Criteria:

* IHCA (unwitnessed IHCA with initial asystole; these patients may still be eligible if visible or audible signs of life were witnessed within 10 minutes after IHCA (no-flow duration ≤10 minutes, in keeping with the non-inclusion criteria for HYPERION study).
* Sustained ROSC (Return Of Spontaneous Circulation) defined as signs of circulation for 20 minutes without chest compressions
* At least 1 mg of epinephrine
* Coma defined as an inability to obey verbal commands (Glasgow Coma Scale motor response <6 or Full Outline of UnResponsiveness (FOUR) score motor response <4) after sustained ROSC
* Eligible for intensive care without restrictions or limitations
* Inclusion within 90 minutes of ROSC
* Age 18 years or older
* Next of kin informed about the trial and having consented to participation of the patient in the trial (patients with coma are unable to consent). If no next of kin can be contacted during screening for the study, trial inclusion will be completed as an emergency procedure by the ICU physician, in compliance with Country of inclusion law.
* Healthcare costs covered by the French statutory healthcare insurance system

Exclusion Criteria:

* Temperature at admission <30°C
* Obvious or suspected pregnancy
* Intracranial bleeding
* Dependent on others for activities of daily living before hospitalization
* Patient under curators, guardianship or under protection of justice
* Correctional facility inmate
* Patient who does no speak French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 788 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
To assess whether induced hypothermia (TTM at 33°C) is superior to targeted normothermia in providing a favorable neurological outcome, defined as a modified Rankin Scale (mRS) score of 0 to 3 at 6 months. | 6 months after randomization
  The primary endpoint is a favorable neurological outcome at 6 months, defined as an mRS score between 0 and 3.

SECONDARY OUTCOMES:
All-cause mortality 2 months after randomization | 2 months after randomization
  Causes of death (refractory hemodynamic shock, life-support withdrawal for neurological reasons, life-support withdrawal due to comorbidities, respiratory failure, sudden cardiac death, brain death)
All-cause mortality 3 months after randomization | 3 months after randomization
  Causes of death (refractory hemodynamic shock, life-support withdrawal for neurological reasons, life-support withdrawal due to comorbidities, respiratory failure, sudden cardiac death, brain death)
All-cause mortality 4 months after randomization | 4 months after randomization
  Causes of death (refractory hemodynamic shock, life-support withdrawal for neurological reasons, life-support withdrawal due to comorbidities, respiratory failure, sudden cardiac death, brain death)
All-cause mortality 6 months after randomization | 6 months after randomization
  Causes of death (refractory hemodynamic shock, life-support withdrawal for neurological reasons, life-support withdrawal due to comorbidities, respiratory failure, sudden cardiac death, brain death)
ICU lengths of stay | from day of randomization until the day of discharge from ICU, an average of 20 days.
Hospital lengths stay | from day of randomization until the day of discharge from hospital, an average of 20 days.
Neurological outcome measured by modified Rankin Scale (mRS) score, ranging from 0 to 6 at 2 months after randomization | 2 months after randomization
Neurological outcome measured by modified Rankin Scale (mRS) score, ranging from 0 to 6 at 3 months after randomization | 3 months after randomization
  A score of 0 to 3 is considered a favorable neurological outcome.
Neurological outcome measured by modified Rankin Scale (mRS) score ranging from 0 to 6 at 4 months after randomization | 4 months after randomization
  A score of 0 to 3 is considered a favorable neurological outcome.
Mechanical ventilation duration | from time of randomization to final extubation or up to 28 days
  A score of 0 to 3 is considered a favorable neurological outcome.
Biomarkers concentration : neuron-specific enolase (NSE) on day 0 | at day 0
Biomarkers concentration : neuron-specific enolase (NSE) on day 2 | at day 2
Biomarkers concentration : neuron-specific enolase (NSE) on day 3 | at day 3
Biomarkers concentration : neurofilament light chain (NFL) on day 2 | at day 2
Health-related quality of life (HRQoL) assessed using the 36-item Short Form Health Survey (SF-36) 6 months after randomization | 6 months after randomization
Cognitive dysfunction assessed using the Montreal Cognitive Assessment (MoCA) 6 months after randomization | 6 months after randomization
Complications during ICU stay : nosocomial infections | from day of randomization until the day of discharge from ICU, or up to 28 days.
Complications during ICU stay : severe arrhythmias | from day of randomization until the day of discharge from ICU, or up to 28 days.
Complications during ICU stay : venous thromboembolism | from day of randomization until the day of discharge from ICU, or up to 28 days.
Complications during ICU stay : ischemic complications | from day of randomization until the day of discharge from ICU, or up to 28 days.
Complications during ICU stay : sedations complications | from day of randomization until the day of discharge from ICU, or up to 28 days.

CONTACTS AND LOCATIONS:
Locations (32):
- Belgium (5):
  - Hôpital Erasme, Brussels
  - CHU Charleroi, Charleroi
  - Hôpital Universitaire de Gand, Ghent
  - Hôpital Universitaire de Bruxelles, Jette
  - Clinique Saint-PIerre, Ottignies
- France (26):
  - CH d'Angoulême, Angoulême
  - CH Dubois Brive, Brive-la-Gaillarde
  - CHU de Caen, Caen
  - Hôpital Simone Veil, Cannes
  - CH Public du Cotentin, Cherbourg
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Bocage, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - Hôpital André Mignot, Le Chesnay
  - CHRU- Hôpital Roger Salengro, Lille
  - CHU Dupuytren, Limoges
  - Hôpital Edouard Herriot, Lyon
  - APHM - Hôpital Nord, Marseille
  - Hôpital Privé Jacques Cartier, Massy
  - CHU de Nantes, Nantes
  - Hôpital de l'Archet, Nice
  - CHR d'Orléans, Orléans
  - APHP-Hôpital Saint-Antoine, Paris
  - APHP- Hôpital Cochin, Paris
  - APHP - Hôpital Ambroise Paré, Paris
  - CH de Roanne, Roanne
  - CH de Rodez, Rodez
  - CHRU de Strasbourg, Strasbourg
  - Hôpital Sainte-Musse, Toulon
  - CHRU de Tours, Tours
  - CH Brocéliande Atlantique, Vannes
- CHU Les Abymes, Pointe-à-Pitre, La Guadeloupe, Guadeloupe